CLINICAL TRIAL: NCT00761748
Title: A Comparative, Randomised, Crossover Study With SenSura Uro 2-piece Versus ConvaTec 2-piece Among 30 Urostomy-operated Persons in Germany
Brief Title: Comparison of Two Urostomy Bags (2-piece).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DK189OS
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Results first posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-11

CONDITIONS: Urostomy Patent
Keywords: Urostomy,; 2-piece,; preference,

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SenSura (Experimental): SenSura Uro 2-piece. Is a urostomy bag with the intended use of collecting urine from a stoma. Consist of a base plate and a bag that is attached to the base plate.
  Interventions: Device: SenSura Uro 2-piece
- Convatec (Active Comparator): Convatec Uro 2-piece Is a urostomy bag with the intended use of collecting urine from a stoma. Consist of a base plate and a bag that is attached to the base plate.
  Interventions: Device: Convatec Uro 2-piece

INTERVENTIONS:
Device: Convatec Uro 2-piece — Specific name of the device: 'Combihesive Natura® with a Durahesive Convex-It® base plate, 45 mm coupling, moldable (13-22 and 22-33 mm) hole size with boarder tape'.
  The subjects are asked to test each of the two products for 21 days plus/minus 3 days in a randomised order and in accordance with their normal frequency of change and normal use pattern. The duration of the clinical investigation should be enough time to identify any difference in user-preference. If the subject is in the middle of testing an urostomy base plate when the test period is turning into the next period, the urostomy base plate can be worn until it needs to be changed. It is not possible to blind the investigation as the appearance of the test- and refer-ence products are very different in the look.
  Other Names: ConvaTec 2-piece
  Arms: Convatec
Device: SenSura Uro 2-piece — SenSura URO 2-piece Extended Wear, convex light, 50 mm coupling, cuttable (15-33 mm)
  Other Names: SenSura
  Arms: SenSura

SUMMARY:
Coloplast A/S has developed a new, improved 2-piece product for people with urostomies.

DETAILED DESCRIPTION:
The 2-piece product is a part of a new product family, under the brand name SenSura. The aim of this investigation is to see how the urology product is perceived and how it performs against another 2-piece product from ConvaTec. The device 'ConvaTec 2-piece combihesive Natura' is selected as the comparative product because of its similarity to SenSura 2-piece product.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old,
* Be able to complete a written consent form
* Be able to fill in the Case Report Form
* Have a urostomy with a diameter of 33 mm. or less.
* Have had the urostomy for 3 months or more.
* Use a 2-piece convex (or convex light) normally.
* Be able to use SenSura URO 2-piece product
* Be able to use ConvaTec, 2-piece product
* Be able to handle the product themselves (application, removal and emptying),

Exclusion Criteria:

* In order to be enrolled in the clinical investigation, the subjects must not:

  * Need to use an ostomy belt
  * Be currently suffering from any dermatological problems, needing special treatment, on the peristomal skin
  * Being treated with chemo- or radiation therapy,
  * Be hospitalized during study enrollment, or have a hospitalization or significant surgery planned during the 4-week study period, or
  * Be pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Carter, M.Sc, Study Chair — Coloplast A/S
Locations (1):
- Visé Mitteldeutschland GmbH, Magdeburg, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were recruited by the investigators at multiple sites in Germany.
Pre-assignment Details: 39 subjects were enrolled in the study, however 9 subjects were excluded from participating in the study.
Groups:
- Sensura Uro 2 Piece First, Then Convatec 2 Piece: Sensura is a newly developed two piece product for people with urostomies.
- ConvaTec 2 Piece,First, Then Sensura Uro 2 Piece: Convatec is the reference product and was chosen because of its similarity with the Sensura appliance.
Period: First Intervention (21 +/- 3 Days)
Arm/Group | Sensura Uro 2 Piece First, Then Convatec 2 Piece | ConvaTec 2 Piece,First, Then Sensura Uro 2 Piece
Started | 20 | 10
Completed | 17 | 7
Not Completed | 3 | 3
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 0 | 3
Period: Second Intervention (21 +/- 3 Days)
Arm/Group | Sensura Uro 2 Piece First, Then Convatec 2 Piece | ConvaTec 2 Piece,First, Then Sensura Uro 2 Piece
Started | 17 | 7
Completed | 17 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: Urostomy operated subjects
Arm/Group | Overall Study Population
Number analyzed (Participants) | 30
Age Continuous [Median (Full Range); unit: years] | 68 [42 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Preference of the Two Urostomy Products
Description: Number of participants preferring the SenSura Uro 2 piece product or the reference Convatec 2 piece product.
  The subjects are asked via the case report form (questionnaire) at the end of the second cross over period, which of the two products they preferred.
Time Frame: 6 weeks
Population: The Per protocol (PP) population is analysed. PP-criteria: Subjects fulfill the inclusion and exclusion criteria, do not seriously violate the protocol, are exposed to both products and are evaluable with respect to the primary endpoint (state preference). *One drop out was evaluable, as the subject tried both products and stated a preference.
Measure: Number; unit: participants
Groups:
- Sensura Uro 2 Piece: The new SenSura Uro 2-piece. Is a urostomy bag with the intended use of collecting urine from a stoma. Consist of a base plate and a bag that is attached to the base plate.
- Convatec 2 Piece: The reference product Convatec 2 piece is a urostomy bag intended for collecting urin from a stoma.
Arm/Group | Sensura Uro 2 Piece | Convatec 2 Piece
Number analyzed (Participants) | 25 | 25
participants | 21 | 4

ADVERSE EVENTS:
Groups:
- Sensura Uro 2 Piece: SenSura Uro 2-piece. Is a urostomy bag with the intended use of collecting urine from a stoma. Consist of a base plate and a bag that is attached to the base plate.
- Convatec 2 Piece: The reference product Convatec 2 piece is a urostomy bag intended for collecting urine from a stoma.
Arm/Group | Sensura Uro 2 Piece | Convatec 2 Piece
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30
Other Adverse Events (participants affected / at risk) | 5/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensura Uro 2 Piece (N=30) | Convatec 2 Piece (N=30)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensura Uro 2 Piece (N=30) | Convatec 2 Piece (N=30)
Skin irritation (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less